CLINICAL TRIAL: NCT06857448
Title: Autologous Point-of-Care Adipose Therapy for Reconstruction and Regeneration of Traumatized Skin: Recent Injury
Brief Title: Autologous Point-of-Care Adipose Therapy: Recent Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Armed Forces Institute of Regenerative Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Francesco Egro, Director of Burn Reconstruction, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY24080150 - Recent Injury
Record Dates: First submitted 2025-02-04; First posted 2025-03-04 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Burns; Contracture Scar; Surgical Injury
Keywords: fasciotomy; trauma
MeSH Terms: conditions — Burns; Intraoperative Complications; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Autologous Layered Composite Grafting consists of the layered strategy of simultaneous fat and skin grafting. Fat is harvested by minimally invasive liposuction and applied directly to the wound base without any chemical or biologic processing. Skin is harvested as per standard of care and applied either to the wound bed directly as per controls or to the layer of adipose tissue.
  Investigators will compare quality of acute reconstruction across two treatment arms after fasciotomy, trauma and/or burn defects (68 subjects).
  * Group 1: Split Thickness Skin Graft (STSG) Reconstruction;
  * Group 2: Base of wound fat graft with STSG Reconstruction (Autologous Layered Composite Grafting).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Split Thickness Skin Graft (STSG) Reconstruction (Active Comparator): In this Arm, the investigators will evaluate full thickness defects generated after fasciotomy, trauma debridement, and/or burn excision of the face, neck, or extremities. These wounds represent common, full-thickness injuries, which require prolonged recovery and dressing changes as bridge to either skin graft or delayed closure and commonly are associated with contour irregularities, adhesions, and contracture. The investigators will assess current standard of care dressing changes followed by immediate STSG.
  Interventions: Procedure: Split Thickness Skin Graft (STSG)
- Base of wound fat graft with STSG Reconstruction (Autologous Layered Composite Grafting). (Experimental): In this Arm, the investigators will evaluate full thickness defects generated after fasciotomy, trauma debridement, and/or burn excision of the face, neck, or extremities. These wounds represent common, full-thickness injuries, which require prolonged recovery and dressing changes as bridge to either skin graft or delayed closure and commonly are associated with contour irregularities, adhesions, and contracture. The investigators will assess current standard of care dressing changes followed by base of wound fat graft with STSG reconstruction (Autologous Layered Composite Grafting).
  Interventions: Procedure: Base of wound fat graft with STSG Reconstruction (Autologous Layered Composite Grafting).

INTERVENTIONS:
Procedure: Split Thickness Skin Graft (STSG) — Partial thickness skin in STSGs are performed by harvesting via dermatome the donor site. Donor sites are typically taken from a flat surface on the thigh, lower back, or gluteal region to allow for a graft of even thickness and the selection of donor site is to be based on clinical standard practice. These grafts are placed on the prepared recipient site.
  Arms: Acute Split Thickness Skin Graft (STSG) Reconstruction
Procedure: Base of wound fat graft with STSG Reconstruction (Autologous Layered Composite Grafting). — Autologous Layered Composite Grafting consists of the layered strategy of simultaneous fat and skin grafting. Fat is harvested by minimally invasive liposuction and applied directly to the wound base without any chemical or biologic processing. Skin is harvested as a split thickness skin graft by dermatome and applied over the layer of adipose tissue.
  Arms: Base of wound fat graft with STSG Reconstruction (Autologous Layered Composite Grafting).

SUMMARY:
The goal of this study is to explore if an adipose-based therapeutic strategy can treat full-thickness soft-tissue trauma wounds in injured individuals, especially those with severe burns or soft-tissue loss. The main question it aims to answer are:

- Can immediate autologous adipose and autologous layered composite grafting be effective for acute functional soft-tissue reconstruction?

Researchers will compare the single-stage autologous layered composite grafting method to traditional methods to see if it improves healing outcomes, minimizes scarring, and reduces infection risk.

Participants will:

* Receive immediate fat grafting into the wound.
* Undergo simultaneous split-thickness skin grafting for full soft-tissue reconstruction.

DETAILED DESCRIPTION:
Soft-tissue injuries from blasts, burns, or multiple traumas can cause severe damage, leading to loss of function, lower quality of life, long recovery times, and inability to work. When these injuries involve deep burns or full-thickness tissue loss in areas that move a lot, they are especially difficult to treat due to the risk of scarring, stiffness, and tissue sticking together. There is a need for a reliable, single-stage treatment that can provide soft, flexible tissue reconstruction with minimal risk, cost, and, complexity. To address this issue, the investigators propose a fat-based approach to reconstruction. Fat tissue is easily available from the patient's own body and carries many benefits in reconstructive surgery. Our team has shown that using a layer of fat immediately in treatment creates a soft, vascular layer that reduces scarring, improves tissue volume, and supports a one-stage, multi-layer reconstruction without the need for complex surgery or causing harm to the donor area. The purpose of this study is to compare this reconstructive approach under the following conditions:

• Demonstrate efficacy of immediate autologous adipose and autologous layered Composite Grafting in acute functional soft-tissue reconstruction.

Evaluators including dedicated observers will be blinded to treatment group/strategy.

ELIGIBILITY:
Inclusion Criteria:

* The proposed study will include adult patients 18 years of age or older,
* male or female,
* civilian, military, active duty or retired veterans
* presenting for unilateral or bilateral fasciotomy of the extremity at any level necessary
* secondary to non-infectious etiology,
* unilateral or bilateral traumatic full-thickness skin loss of the face, head, neck or extremities necessitating reconstruction, and/or
* full or partial thickness burn injury of the face, neck, or extremity requiring excision and/or reconstruction.
* Additional inclusion criteria includes willingness to be randomized to receive a fat graft.

Exclusion Criteria:

* Age < 18 years of age,
* active infection,
* medical co-morbidities or anatomic configuration deemed by the physician to be a concern for safety,
* unwilling or unable to comply with study procedures,
* radiation to the site of interest,
* prisoners and/or vulnerable populations.
* In addition, candidates that are pregnant or plan to become pregnant in the next year, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Total score on the Patient and Observer Scar Assessment Scale (POSAS): Pigmentation, Pliability, Vascularity, Thickness, Relief, and Surface Area, collected at the 9 month follow up visit. | From surgery to 9-month clinical endpoint.
  POSAS measures subjective assessment on a 1-10 scale from normal skin to worst scar imaginable across 6 metrics (surface area, vascularity, pigmentation, thickness, pliability and relief). The lowest sum score, reflecting normal skin, is 6 and the highest score, reflecting the worst imaginable scar, is 60.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability). | From surgery to 9-month clinical endpoint.
  Incidence of adverse events will be reported for all study participants.
Number of Operative Encounters | From surgery to 9-month clinical endpoint.
  The investigators will additionally assess early outcome metrics including number of operative encounters.
Percent Graft Take | From surgery to 9-month clinical endpoint.
  The investigators will additionally assess early outcome metrics including percent graft take (% of surface area).
Time to Final Healing/Graft Take | From surgery to 9-month clinical endpoint.
  The investigators will additionally assess early outcome metrics including, time to final healing/graft take in days.
Photographic Appearance of Wound | From surgery to 9-month clinical endpoint.
  Photographic evaluation for wound appearance. This is gross appearance.
Area of Wound | From surgery to 9-month clinical endpoint.
  Photographic evaluation for size of wound area. This is measured in cm2
Tissue Thickness | From surgery to 9-month clinical endpoint.
  The investigators will measure tissue thickness as determined by ultrasound.
Pliability (Tensiometry/Cutometry) | From surgery to 9-month clinical endpoint.
  The investigators will utilize a noninvasive cutometer/tensiometer to determine tissue pliability.
Tissue Mobility (Resistance to Adhesion) | From surgery to 9-month clinical endpoint.
  The investigators will measure tissue mobility under non-invasive tissue stretch. Measurement is achieved by the mm of stretch achievable from a given point under a standardized stress.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Egro, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Mercy Hospital, Pittsburgh, Pennsylvania
  - Presbyterian Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piccolo NS, Piccolo MS, Piccolo MT. Fat grafting for treatment of burns, burn scars, and other difficult wounds. Clin Plast Surg. 2015 Apr;42(2):263-83. doi: 10.1016/j.cps.2014.12.009. Epub 2015 Feb 21. PMID 25827568
- [Background] Simonacci F, Bertozzi N, Grieco MP, Grignaffini E, Raposio E. Procedure, applications, and outcomes of autologous fat grafting. Ann Med Surg (Lond). 2017 Jun 27;20:49-60. doi: 10.1016/j.amsu.2017.06.059. eCollection 2017 Aug. PMID 28702187
- [Background] Evans BGA, Gronet EM, Saint-Cyr MH. How Fat Grafting Works. Plast Reconstr Surg Glob Open. 2020 Jul 14;8(7):e2705. doi: 10.1097/GOX.0000000000002705. eCollection 2020 Jul. PMID 32802628
- [Background] Woodruff SI, Galarneau MR, McCabe CT, Sack DI, Clouser MC. Health-related quality of life among US military personnel injured in combat: findings from the Wounded Warrior Recovery Project. Qual Life Res. 2018 May;27(5):1393-1402. doi: 10.1007/s11136-018-1806-7. Epub 2018 Feb 15. PMID 29450855
- [Background] Mokos ZB, Jovic A, Grgurevic L, Dumic-Cule I, Kostovic K, Ceovic R, Marinovic B. Current Therapeutic Approach to Hypertrophic Scars. Front Med (Lausanne). 2017 Jun 20;4:83. doi: 10.3389/fmed.2017.00083. eCollection 2017. PMID 28676850
- [Background] Finnerty CC, Jeschke MG, Branski LK, Barret JP, Dziewulski P, Herndon DN. Hypertrophic scarring: the greatest unmet challenge after burn injury. Lancet. 2016 Oct 1;388(10052):1427-1436. doi: 10.1016/S0140-6736(16)31406-4. PMID 27707499
- [Background] Marshall CD, Hu MS, Leavitt T, Barnes LA, Lorenz HP, Longaker MT. Cutaneous Scarring: Basic Science, Current Treatments, and Future Directions. Adv Wound Care (New Rochelle). 2018 Feb 1;7(2):29-45. doi: 10.1089/wound.2016.0696. PMID 29392092
- [Background] Wolf JM, Athwal GS, Shin AY, Dennison DG. Acute trauma to the upper extremity: what to do and when to do it. Instr Course Lect. 2010;59:525-38. PMID 20415403
- [Background] Harrison BL, Lakhiani C, Lee MR, Saint-Cyr M. Timing of traumatic upper extremity free flap reconstruction: a systematic review and progress report. Plast Reconstr Surg. 2013 Sep;132(3):591-596. doi: 10.1097/PRS.0b013e31829ad012. PMID 23676968
- [Background] Le TD, Gurney JM, Nnamani NS, Gross KR, Chung KK, Stockinger ZT, Nessen SC, Pusateri AE, Akers KS. A 12-Year Analysis of Nonbattle Injury Among US Service Members Deployed to Iraq and Afghanistan. JAMA Surg. 2018 Sep 1;153(9):800-807. doi: 10.1001/jamasurg.2018.1166. PMID 29847675
- [Background] D'Souza EW, MacGregor AJ, Dougherty AL, Olson AS, Champion HR, Galarneau MR. Combat injury profiles among U.S. military personnel who survived serious wounds in Iraq and Afghanistan: A latent class analysis. PLoS One. 2022 Apr 6;17(4):e0266588. doi: 10.1371/journal.pone.0266588. eCollection 2022. PMID 35385552